CLINICAL TRIAL: NCT06424704
Title: Microbiology of Chronic Suppurative Otitis Media: Prospective Study
Brief Title: Chronic Suppurative Otitis Media Microbiology
Status: Not yet recruiting | Type: Observational
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Bulent Ulusoy, Selcuk University Faculty of Medicine, Selcuk University
Other Study IDs: 2024/145
Record Dates: First submitted 2024-05-16; First posted 2024-05-22 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: Otitis Media, Suppurative Chronic; Cholesteatoma; Microbial Colonization
Keywords: Chronic suppurative otitis media; Cholesteatoma; Ear discharge
MeSH Terms: conditions — Otitis Media; Cholesteatoma; Communicable Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples Without DNA — Culture samples taken from the ears of patients with chronic suppurative otitis media with cholesteatoma and chronic suppurative otitis media without cholesteatom.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Chronic suppurative otitis media with cholesteatoma (Chole): Patients who applied to Selçuk University Faculty of Medicine Hospital, Department of Ear, Nose and Throat Diseases & Head and Neck Surgery with complaints of ear discharge and were diagnosed with chronic suppurative otitis media with cholesteatoma were included in the study.
  Interventions: Diagnostic Test: Microbiological culture
- Chronic suppurative otitis media without cholesteatoma (CSOM): The study included patients who applied to Selçuk University Faculty of Medicine Hospital, Department of Ear, Nose and Throat Diseases & Head and Neck Surgery, with complaints of ear discharge and were diagnosed with chronic suppurative otitis media without cholesteatoma.
  Interventions: Diagnostic Test: Microbiological culture

INTERVENTIONS:
Diagnostic Test: Microbiological culture — Samples taken from chronic suppurative otitis media patients in the Medical Microbiology Laboratory of Selçuk University Faculty of Medicine will be planted in 5% sheep blood Columbia agar, eosin methylene blue agar and saboraud dextrose agar, and the media will be incubated at 37oC for 24-48 hours. Growing bacteria and fungi were examined using traditional methods [Gram staining, catalase test, coagulase test, bacitracin disk, PYR test (L-pyrrolidonyl-β-naphthylamide), oxidase test, IMViC test, lactophenol cotton blue, etc.] and VITEK 2 (bioMerieux, France).
  Other Names: Antibiotic susceptibility tests will be performed with the Kirby Bauer disc diffusion test and VITEK2 automated system (bioMerieux, France).

SUMMARY:
This study is planned to reveal the microbiological agents and drug sensitivities to these agents in patients diagnosed with chronic suppurative otitis media who complain of ear discharge.

DETAILED DESCRIPTION:
Patients with complaints of ear discharge and who were diagnosed with chronic suppurative otitis media will be included in the study. Patients will be divided into two groups: CSOM with cholesteatoma and CSOM without cholesteatoma. One hundred ten patients from each group will be included in the study. After a comprehensive medical history is taken for each patient, the patient's external auditory canal will be cleaned with sterile aspirators. A sterile culture will be taken from the discharge of the ear and sent to microbiology. With the data obtained from microbiological examination, pathogens will be classified as gram-positive, gram-negative, anaerobic, and fungal and examined according to monomicrobial and polymicrobial growth. Antibiotic susceptibility tests will be conducted to determine the effectiveness of antibiotics against the bacteria causing the infection.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with chronic suppurative otitis media
2. Patients over 18 years of age

Exclusion Criteria:

1. Chronic nonsuppurative otitis media patients
2. Patients diagnosed with external ear canal/middle ear malignancy
3. Patients who take immunosuppressive drugs
4. Immunosuppressive patients
5. Patients who used antibiotics (topical-systemic) in the last week

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will include patients who applied to Selçuk University Faculty of Medicine Hospital, Department of Ear, Nose and Throat Diseases & Head and Neck Surgery, with complaints of ear discharge and were diagnosed with chronic suppurative otitis media.
Sampling Method: Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2024-05-15 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Microbiology of chronic suppurative otitis media | 2024-2026 (24 months)
  Microbiology in patients diagnosed with chronic suppurative otitis media with and without cholesteatoma

SECONDARY OUTCOMES:
Antibiotic susceptibility in chronic suppurative otitis media | 2024-2026 (24 months)
  Investigation of antibiotic susceptibility and resistance in patients diagnosed with chronic suppurative otitis media with and without cholesteatoma.

CONTACTS AND LOCATIONS:
Overall Officials: Bulent Ulusoy, MD, Principal Investigator — Selcuk University
Locations (2):
- Turkey (Türkiye) (2):
  - Bulent ULUSOY, Konya, Selcuklu
  - Selcuk University, Konya, Selcuklu

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Khairkar M, Deshmukh P, Maity H, Deotale V. Chronic Suppurative Otitis Media: A Comprehensive Review of Epidemiology, Pathogenesis, Microbiology, and Complications. Cureus. 2023 Aug 18;15(8):e43729. doi: 10.7759/cureus.43729. eCollection 2023 Aug. PMID 37727177
- [Background] Verhoeff M, van der Veen EL, Rovers MM, Sanders EA, Schilder AG. Chronic suppurative otitis media: a review. Int J Pediatr Otorhinolaryngol. 2006 Jan;70(1):1-12. doi: 10.1016/j.ijporl.2005.08.021. Epub 2005 Sep 27. PMID 16198004